CLINICAL TRIAL: NCT07049367
Title: Finger Extension and Tripod Grip as Indicators of Hand Function Improvement in Subacute Stroke Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: DPT/Batch-Fall20/1013
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hand Function Improvement
  Interventions: Diagnostic Test: Hand Function Improvement

INTERVENTIONS:
Diagnostic Test: Hand Function Improvement — Finger Extension and Tripod Grip as Indicators of Hand Function Improvement in Subacute Stroke Patients

SUMMARY:
Finger Extension and Tripod Grip as Indicators of Hand Function Improvement in Subacute Stroke Patients This is a Study design will be Cross Sectional Study Data will be collected from Shadman Medical Center Lahore

ELIGIBILITY:
Inclusion Criteria:

* 40-85 Years of age
* Gender both male and female
* Ischemic stroke, unilateral, first-time stroke
* Impaired sensory-motor function in the upper Limb

Exclusion Criteria:

* Transient ischemic attack
* Other neurological diseases (Parkinson's disease, multiple sclerosis), Hemineglect, no sitting balance
* Co-morbidities

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross-sectional Study on Finger Extension and Tripod Grip as Indicators of Hand Function Improvement in Subacute Stroke Patients
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Nine Hole Peg Test (9-HPT) | 6 Month
  The Nine Hole Peg Test (9-HPT) is a standardized assessment used to evaluate fine motor dexterity and coordination, particularly in individuals with neurological conditions like stroke, multiple sclerosis, or Parkinson's disease. The test involves placing and removing nine pegs into holes on a board as quickly as possible, using one hand at a time. The time taken to complete the task is recorded, and the average of multiple trials is used to assess hand function

CONTACTS AND LOCATIONS:
Locations (1):
- Shadman Medical Center Department of Neurological and Functional Rehabilitation, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No